CLINICAL TRIAL: NCT07070778
Title: The Effect of Upper Extremity Aerobic Exercise Training on Arterial Stiffness in Individuals With Breast Cancer
Brief Title: Arterial Stiffness in Individuals With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/5-39
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Aerobic Exercise; Breast Cancer; Arterial Stiffness
Keywords: breast cancer; Aerobic exercise training; Arterial Stiffness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study consists of one group: this group performs upper extremity aerobic exercise training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper Extremity Aerobic Exercise (Other): Participants will only receive a 12-week upper extremity aerobic exercise training program.
  Interventions: Other: Upper Extremity Aerobic Exercise Training Program

INTERVENTIONS:
Other: Upper Extremity Aerobic Exercise Training Program — 12 weeks of supervised upper limb aerobic exercise training, 3 sessions per week, 25 minutes per session.

SUMMARY:
The aim of this study was to evaluate vascular toxicity induced by anthracyclines and other anticancer drugs and to measure arterial stiffness in women with breast cancer and, in addition, to evaluate the acute and chronic arterial stiffness responses of upper extremity aerobic exercise training.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women both in the world and in our country. Today, with the technological developments, breast cancer treatments have improved considerably and the mortality rate has decreased. However, despite the developments in treatments, the quality of life of patients has still not reached the desired level. Upper extremity dysfunctions are frequently observed in patients after breast cancer treatment. This upper extremity dysfunction causes a decrease in the quality of daily life of patients. Arterial stiffness contributes to hypertension and increases the risk of cardiovascular disease. The American College of Sports Medicine (ACSM) recommends that healthy adults perform moderate to vigorous intensity aerobic exercise at least 5 times per week and resistance exercise 2-3 times per week. Aerobic exercise can reduce arterial stiffness after both acute and chronic interventions. A small number of studies on aerobic exercise have reported that this exercise training improves the functional level of patients after breast cancer. However, the effect of aerobic exercise training on arm exercise capacity and arterial stiffness in patients with breast cancer is still unclear. Thus, the results of this study may guide physiotherapists working in this field about upper extremity exercise training after breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 40-69,
* Baseline left ventricular ejection fraction (LVEF) >50%,
* Absence of coronary artery disease and haemodynamically significant valvular heart disease,
* Absence of carotid atherosclerotic plaques,
* Volunteering to participate in the research,
* At least 15 months after breast cancer surgery,
* No problems in reading and/or understanding the scales and being able to co-operate with the tests.
* Physically inactive (60 minutes of structured exercise per week <).

Exclusion Criteria:

* Presence of active infection,
* Presence of bilateral breast cancer,
* History of surgical, neurological or orthopaedic problems that may affect upper extremity functionality other than breast cancer surgery,
* Having a neurological disease or other clinical diagnosis that may affect cognitive status,
* Left ventricular dysfunction and severe liver and kidney dysfunction before starting chemotherapy
* Musculoskeletal and neurological disease that may affect exercise performance, symptomatic heart disease, previous lung surgery and malignant disease.
* Presence of unstable hypertension or diabetes mellitus.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Arterial Stiffness | one years
  Arterial stiffness will be assessed noninvasively using the pulse wave velocity (PWV) technique with the Mobil-O-GRAPH (TG) (I.E.M., Stolberg, Germany), an oscillometer-based device. Pulse wave velocity, augmentation pressure, reflection magnitude, agumentation index parameters will be recorded.

SECONDARY OUTCOMES:
Comorbidity Assessment | one year
  The Charlson Comorbidity Index According to this index developed by the Institute of Medicine, comorbid diseases are assessed according to their severity. is scored. Comorbidities are scored from mild disease state to severe disease state. are given a score of 1, 2, 3, 4, respectively, and the score obtained by summing the scores of comorbid diseases The severity of comorbidity is also calculated according to the weighted score. One point for every ten years over the age of forty (50-59: 1 point, 60-69: 2 points, etc.)
Maximal Arm Exercise Capacity | one year
  VO2peak requirement during arm ergometry will be estimated using MET levels calculated at each power output based on gender at various body weights and will be displayed in ml/kg/min (1 MET = 3.5 ml/kg/min)
Cardiovascular Disease Risk Scoring | one year
  To be evaluated with SCORE2. The risk calculated according to the SCORE system is accepted as low risk if <1%, medium risk if 1-4%, high risk if 5-9%, and very high risk if 10% and above (16). According to the SCORE2 system, <2.5% is considered low-moderate risk, 2.5%-7.5% is considered high risk, and 7.5% and above is considered very high risk in patients aged <50 years. In those over 50 years of age, <5% is considered low-moderate risk, 5-10% is considered high risk, and 10% and above is considered very high risk.

CONTACTS AND LOCATIONS:
Overall Officials: Melda Saglam, PhD, Study Chair — Hacettepe University; Ebru Calik Kutukcu, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No